CLINICAL TRIAL: NCT01117298
Title: A Randomized Control Trial to Assess the Efficacy of Tadalafil in Raynaud's Phenomenon in Scleroderma: A Double Blind, Parallel Group, Multicentric Study
Brief Title: A Randomized Control Trial to Assess the Efficacy of Tadalafil in Raynaud's Phenomenon in Scleroderma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Collaborators: Institute of Postgraduate Medical Education and Research (Ambiguous); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Army Hospital Research And Referral, India (Other)
Responsible Party: Dr VIkas Agarwal, PI, SGPGIMS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B22:A15:PGI/DM/EC/40/7.11.2007
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Raynaud's Phenomenon; Digital Ulcers; Scleroderma
Keywords: Raynaud's phenomenon; ischemic ulcers; digital ulcers; digital infarcts; gangrene; vasodilators; endothelial dysfunction; scleroderma
MeSH Terms: conditions — Raynaud Disease; digital ulcers; Scleroderma, Diffuse; Gangrene | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental)
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tab Tadalafil, 20 mg alternate day for 8 weeks
  Other Names: Tadalis
  Arms: Tadalafil
Drug: Placebo — Tab Placebo every alternate day for 8 weeks
  Arms: Placebo

SUMMARY:
Raynaud's phenomenon (RP) associated with scleroderma is a difficult problem to treat. Many patients develop ischemic digital ulcers due to severe RP that causes considerable morbidity and adversely affects the quality of life. In an earlier study, we have observed marked improvement in RP attacks and rapid healing of digital ulcers following therapy with phosphodiesterase V inhibitor, Tadalafil. In the present multicentric study we aim to study the efficacy of Tadalafil in patients continuing to have RP attacks despite using at least one or more vasodilators.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects between the ages of 18 years and 65 years will be selected for the study if they have a clinical diagnosis of Raynaud's phenomenon secondary to systemic sclerosis (scleroderma) despite being on vasodilator therapy. Raynaud's phenomenon is defined as a history of cold sensitivity associated with colour changes of cyanosis or pallor. Patients with a history of at least 4 attacks per week during two-week pre-trial period even with treatment with other vasodilators will be recruited. Patients fulfilling the diagnostic criteria of scleroderma (as per American College of Rheumatology criteria) or having presence of at least 3 of the 5 features of the CREST syndrome (calcinosis, Raynaud's phenomenon, esophageal dysmotility, sclerodactyly, telangiectasias)will be invited to participate in the study.

Exclusion Criteria:

Patients with:

* Symptomatic orthostatic hypotension,
* Evidence of current malignancy,
* History of sympathectomy,
* Upper extremity deep vein thrombosis or lymphedema within 3 months,
* Recent surgical procedure requiring general anesthesia,
* Acute Myocardial Infarction, unstable angina, strokes and transient ischemic attacks within the past three months,
* Smoking,
* Use of any investigational drug within 30 days of the study sessions,
* Use of medications that might interfere with tadalafil like nitrates and alpha adrenergic blockers that have vasoactive effects, and patients taking potent inhibitors of CYP3A4 such as ritonavir, ketoconazole, and itraconazole, erythromycin, itraconazole, and grapefruit juice,
* Patients taking alcohol,
* Patients with bleeding disorders
* Significant active peptic ulceration,
* Current pregnancy,
* Current breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Daily frequency, duration and severity of Raynaud's phenomenon | Baseline and 8 weeks
Appearance or healing of digital ulcers | Baseline and 8 weeks

SECONDARY OUTCOMES:
Improvement in health assessment questionnaire | Baseline and 8 weeks
Improvement in scleroderma specific health assessment questionnaire | Baseline and 8 weeks
Improvement in quality of life | Baseline and 8 weeks
Improvement in biomarkers of endothelial dysfunction | Baseline and 8 weeks
Improvement in flow mediated dilatation | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Parasar Ghosh, MD, DM, Principal Investigator — IPGMER, Kolkatta; Aman Sharma, MD, Principal Investigator — PGIMER, Chandigarh; Darshan S Bhakuni, MD, Principal Investigator — Army R&R Hospital, New Delhi
Locations (4):
- India (4):
  - Department of Clinical Immunology, Army R&R hospital, New Delhi, ND
  - Medicine Unit II, PGIMER, Chandigarh, Punjab
  - Department of Immunology, SGPGIMS, Lucknow, Uttar Pradesh
  - Immunology Rheumatology Unit, IPGMER, Kolkata, West Bengal

REFERENCES:
- [Derived] Maltez N, Maxwell LJ, Rirash F, Tanjong Ghogomu E, Harding SE, Tingey PC, Wells GA, Tugwell P, Pope J. Phosphodiesterase 5 inhibitors (PDE5i) for the treatment of Raynaud's phenomenon. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD014089. doi: 10.1002/14651858.CD014089. PMID 37929840
- See also: Related Info — http://www.medscape.com/viewarticle/582592